CLINICAL TRIAL: NCT03363061
Title: Prospective Collection of Clinical and Laboratory Variables of Patients Receiving Antithrombotics and Requiring Colonoscopy
Brief Title: Patients on Antithrombotics for Colonoscopy
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Mak Wing Yan, Associate professor, Chinese University of Hong Kong
Other Study IDs: Colon Registry
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Antithrombotics; Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Antithrombotics: The patients should be on antithrombotics on the day of colonoscopy arrangement

SUMMARY:
The use of antithrombotics (antiplatelet agents and anticoagulants) is increasing with an aging global population.Management of antithrombotics in patients undergoing invasive procedures including gastrointestinal endoscopy remains a challenge. Management approach includes taking a precarious balance between the risk of thromboembolism after interruption of antithrombotics and risk of bleeding with the continuation of antithrombotics. Colonoscopy remains one of the commonest endoscopic procedures performed. The optimal management strategy of different antithrombotics during colonoscopy remains unclear.

DETAILED DESCRIPTION:
The use of antithrombotics (antiplatelet agents and anticoagulants) is increasing with an aging global population. Cardiovascular disease is a leading cause of death worldwide. Clinical Practice Research Datalink (CPRD) GOLD database suggests that over 915 000 people in the UK have suffered a myocardial infarction and over 1.3 million are living with angina in 2013. Two percent of people in developed countries are on long-term anticoagulation and up to 10% in the elderly population. Management of antithrombotics in patients undergoing invasive procedures including gastrointestinal endoscopy remains a challenge. Management approach includes taking a precarious balance between the risk of thromboembolism after interruption of antithrombotics and risk of bleeding with the continuation of antithrombotics. The availability of new antithrombotic agents adds to the complexity of antithrombotic management during endoscopy. Warfarin has been the only oral anticoagulant available until the introduction of direct oral anticoagulants (DOACs). Newer antiplatelet agents (prasugrel and ticagrelor, vorapaxar) are becoming more commonly used for the treatment of the acute coronary syndrome.

There remain gaps in the management approach of patients receiving antithrombotics and requiring endoscopy. It is still uncertain of the actual bleeding risk associated with antithrombotic use during endoscopy. Colonoscopy remains one of the commonest endoscopic procedures performed. It is the gold standard for direct evaluation of the colon for patients with the suspected colonic disease. It is also used as a screening test for prevention of colorectal cancer by colonoscopic polypectomy of precancerous polyps.The optimal management strategy of different antithrombotics during colonoscopy remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be over 18 years of age
* Patients undergoing elective colonoscopy for any indication, who are receiving antithrombotics
* Informed consent is obtained

Exclusion Criteria:

* Patients under 18 years of age
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving antithrombotics at colonoscopy arrangement and undergoing elective colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2017-12-08 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Delayed post polypectomy bleeding | Within 30 days
  Delayed post polypectomy bleeding is defined as blood per rectum occurring after colonoscope has been retracted from the anus to 30 days after the procedure requiring hospitalization or treatment.

SECONDARY OUTCOMES:
Immediate post polypectomy bleeding | During Colonoscopy
  Immediate post polypectomy bleeding is defined as bleeding at the time of colonoscopy after polypectomy and requiring endoscopic intervention at the same colonoscopy.
Serious cardiovascular event | Within 6 months.
  Serious cardiovascular event is defined as nonfatal myocardial infarction, nonfatal stroke, or death from a vascular cause as defined by Anti-Platelet Trialists Collaboration criteria within 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Moe Htet Kyaw, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Jiang W, Suen BY, Ho HT, Ching JYL, Chan FKL, Mak JWY. Impact of Physicians' and Patients' Compliance on Outcomes of Colonoscopic Polypectomy With Anti-Thrombotic Therapy. Clin Gastroenterol Hepatol. 2021 Dec;19(12):2559-2566.e1. doi: 10.1016/j.cgh.2020.09.019. Epub 2020 Sep 12. PMID 32931958